CLINICAL TRIAL: NCT03836976
Title: Detection and Amelioration of Gamma Oscillation Abnormalities in Blast-Related Brain Injury
Acronym: DAGABBI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: N3162-P; I21RX003162 (NIH)
Record Dates: First submitted 2019-01-30; First posted 2019-02-11 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: mTBI
Keywords: mild traumatic brain injury; EEG; neuroplasticity; gamma oscillation
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Intervention Model Description: Single arm. All participants will receive auditory gamma-frequency sensory stimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All participants (Experimental): All participants receive auditory gamma sensory stimulation.
  Interventions: Other: Auditory gamma sensory stimulation

INTERVENTIONS:
Other: Auditory gamma sensory stimulation — Gamma-conditioning stimulation will be
  administered in 2 blocks of 3 min each. During each block, participants will be presented with a continuous
  tone at the CF (500 or 1200 Hz) that will be amplitude modulated at 40 H

SUMMARY:
Combat Veterans of post-9/11 conflicts have experienced serious cognitive and emotional problems resulting from exposure to blasts. Recent work suggests that a critical factor influencing the consequences of blast exposure is distance from the blast, rather than the presence or absence of concussion symptoms. Exposure to blasts from a distance of <10 m has been associated with significantly greater cognitive and neural problems than exposure to blasts from >10 m. So far, the effects of blast-related brain injury on the brain are poorly understood, as to date the effects of blast exposure have received little research focus. The investigators propose to use oscillations in the gamma band (30-100 Hz) of the electroencephalogram (EEG; brain waves) to detect and remediate neural circuit dysfunction related to blast injury in Veterans. If successful, this project could lead to new approaches to detect and remediate the effects of blast exposure on Veterans and aid in their functional recovery.

DETAILED DESCRIPTION:
Veterans of recent conflicts have experienced serious cognitive and emotional problems resulting from exposure to blasts. Recent work suggests that a critical factor in the sequelae of blast exposure is distance from the blast, rather than the presence or absence of concussion symptoms. Exposure to blasts from a distance of <10 m has been associated with significantly greater cognitive and neural disturbances than exposure to blasts from >10 m. The neural correlates of blast-related brain injury are poorly understood, as to date this type of brain injury has received little research focus. The investigators propose to use oscillations in the gamma band (30-100 Hz) of the electroencephalogram (EEG) to detect and remediate neural circuit dysfunction related to blast injury in Veterans. Gamma band oscillations have been shown to be involved in several brain functions, including visual perception, selective attention, working memory, long term memory, and motor control. Recent studies in animal models have linked the effects of traumatic brain injury to parvalbumin-expressing (PV+) inhibitory interneurons, which are a critical element of the cortical circuitry that generates gamma oscillations. PV+ interneuron dysfunction is associated with deficits in evoked gamma oscillations and increased power of broadband gamma "noise", as well as cognitive deficits. It has also recently been shown that stimulation of PV+ interneurons by patterned stimuli in the gamma band can improve the function of these interneurons, as well as cognitive function, in animal models of neuropsychiatric disorders. Hence, the investigators believe that gamma oscillations and stimulation provide promising targets for investigation in Veterans who suffer from blast-related brain injury. The investigators will investigate gamma band activity and stimulation in 50 Veterans who will be recruited from the participant pool of the VA Translational Research Center for TBI and Stress Disorders (TRACTS) at the VA Boston Healthcare System.

* Aim 1: To assess whether evoked gamma deficits and increased gamma noise are present in individuals exposed to Close (<10 m) vs. Far (>10 m) blasts. The investigators predict that evoked gamma will be reduced in power and phase synchrony, while gamma noise will be increased in power, in Close compared to Far blast groups.
* Aim 2: To determine whether gamma oscillation abnormalities associated with close blast exposure can be remediated by non-invasive patterned sensory stimulation in the gamma band. The investigators will administer 6 min of auditory steady-state stimulation at 40 Hz. The investigators predict that gamma conditioning will increase evoked gamma oscillations elicited by tones at the conditioned vs. unconditioned frequency, while gamma noise will be decreased. These effects will be greater in the Close compared to the Far blast groups.

This project also has 2 exploratory aims:

* 1) To investigate whether resting state delta-band (1-4 Hz) EEG power is increased in Close relative to Far blast exposure groups, as delta power is increased in individuals who have experienced mild traumatic brain injury compared to healthy controls.
* 2) As blast exposure is associated with white matter deficits, and PV+ interneuron axons are myelinated, the investigators will examine whether gamma abnormalities are correlated with white matter deficits as assessed by diffusion tensor imaging (DTI) measures in the auditory cortex, available from the TRACTS database.

In sum, this project seeks to advance the understanding of the effects of blasts on brain function in Veterans by probing the effects of blast exposure on the neural circuits that generate gamma oscillations, and by testing whether a new type of non-invasive brain stimulation can improve brain function in Veterans exposed to blasts. If successful, this project could lead to new approaches to detect and remediate the effects of blast exposure on Veterans and aid in their functional recovery.

ELIGIBILITY:
Inclusion Criteria:

* Research participants will be 50 veterans
* Ages 18-65 years
* Have experienced blast exposure
* Recruited from the VA Translational Research Center for TBI and Stress Disorders (TRACTS) at the VA Boston Healthcare System (VABHS)
* Half of the participants will have experienced blast exposure from a Close distance (<10 m)
* Half of the participants will have experienced blast exposure from a Far distance (>10 m)
* These groups will be matched on age and female/male ratio

Exclusion Criteria:

Initial exclusion criteria for TRACTS are:

* History of neurological illness

  * Huntington's
  * Parkinson's
  * dementia, etc
* History of seizure disorders unrelated to head injury
* Current diagnosis of schizophrenia, bipolar, or other psychotic disorder
* Self-reported severe depression or anxiety requiring hospitalization overnight, or current active homicidal and/or suicidal ideation with intent requiring crisis intervention
* Cognitive disorder due to general medical condition other than TBI
* Unstable psychological diagnosis (suspected psychotic or personality disorder) that would interfere with accurate data collection, determined by consensus of at least three doctoral-level psychologists.

Additional exclusion criteria for participants in the present project will be:

* Current alcohol or drug dependence, or abuse within the last 6 months (DSM-IV criteria)
* Hearing impairments as assessed by audiometry

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-12-02 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in evoked gamma power of conditioned vs. unconditioned tones | 0 minutes
  Evoked power of the early auditory-evoked gamma oscillation for conditioned vs. unconditioned tones relative to baseline at 0 min after conditioning stimulation.
Change in evoked gamma power of conditioned vs. unconditioned tones | 20 minutes
  Evoked power of the early auditory-evoked gamma oscillation for conditioned vs. unconditioned tones relative to baseline at 20 min after conditioning stimulation.
Change in spontaneous gamma power | 0 minutes
  Spontaneous broadband gamma power relative to baseline at 0 min after conditioning stimulation.
Change in spontaneous gamma power | 20 minutes
  Spontaneous broadband gamma power relative to baseline at 20 min after conditioning stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin M. Spencer, PhD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No